CLINICAL TRIAL: NCT02904798
Title: The Effects of Visible Light on the Skin After Administration of Oral Polypodium Leucotomos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Principle Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#8385
Record Dates: First submitted 2014-06-02; First posted 2016-09-19 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Photodermatoses
Keywords: sunscreen; photoprotection; visible light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polypodium Leucotomos Extract (PLE) (Experimental): Patient will serve as their own control and will be exposed to 4 doses of visible light on one side of their back prior to receiving PLE.
  PLE 240mg will be dispensed to patient after evaluation of Pre-PLE visible light doses are evaluated to be taken by the patient for a total of 28 day followed by exposure of the opposite side of the back with the same 4 doses of visible light as above
  Interventions: Drug: Polypodium Leucotomos

INTERVENTIONS:
Drug: Polypodium Leucotomos — - PL 240mg to be taken by the patient for 28 days prior to irradiation with visible light
  Other Names: Helicocare

SUMMARY:
Polypodium Leucotomos Extract (PLE) is a tropical fern that has antioxidative, photoprotective, chemoprotective, anti-inflammatory, and immunomodulatory properties. The antioxidative effects of PL include inhibition and scavenging of free radicals, lipid peroxidation and reactive oxygen species (ROS) such hydrogen peroxide, superoxide anion, hydroxyl radical and singlet oxygen. Visible light (400-700 nm) causes pigmentation in melanocompetent individuals and induces DNA damage in the human skin through ROS production. The goal of this study is to determine whether the administration of oral PLE has an effect on the development of visible light induced pigmentation.

DETAILED DESCRIPTION:
Polypodium Leucotomos (PL), a tropical fern that is grown in Central America, has been found to contain active compounds that provide antioxidative, photoprotective, chemoprotective, anti-inflammatory, and immunomodulatory properties.The antioxidative effects of PL include inhibition and scavenging of free radicals, lipid peroxidation and reactive oxygen species (ROS) such hydrogen peroxide, superoxide anion, hydroxyl radical and singlet oxygen.Ultraviolet radiation (UVR) and visible light (400-700 nm) can induce DNA damage in the human skin through ROS production.

The visible spectrum is the part of the electromagnetic radiation that is visible to the human eye. While many of the photodermatology studies have focused mainly on the UV portion of the electromagnetic radiation spectrum, as of lately, there have been more studies on visible light. The visible light radiation can exert various biologic effects such as erythema, pigmentation, thermal damage and free radical production. Addtionally, visible light exposure can cause or exacerbate photodermatoses such as solar urticaria, chronic actinic dermatosis (CAD) and cutaneous porphyrias. Sunscreens are the mainstay treatment for these photodermatoses, but often sunscreens offer none to weak protection against visible light.

In the past, studies have studied the erythema development and pigmentary changes induced by visible light. A recent study by Mahmoud et al. reported that visible light induces dark and relatively sustained pigmentation, which has clinical relevance in the treatment of photodermatoses as well as the need for development of filters that protect against visible light.

PURPOSE: To study the effects of visible light on the skin after administration of oral Polypodium leucotomos.

SPECIFIC AIMS:

•Primary objective: Compare the effects of skin irradiated with visible light with and without oral polypodium leucotomos

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 and older
* Patients Fitzpatrick III-VI
* Patient able to understand requirements of the study and risks involved
* Patient able to sign a consent form

Exclusion Criteria:

* A recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation
* A known history of photosensitivity disorders
* A known history of melanoma or non-melanoma skin cancers
* Those planning on going to the tanning parlors
* Using any of the photosensitizing medication
* A woman who is lactating, pregnant, or planning to become pregnant
* Patient planning on exposing the irradiated or control areas to the sun

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-04-23 (Actual)

PRIMARY OUTCOMES:
Difference in pigmentation pre and post administration of oral PLE | 42 days
  Detect differences in visible light induced pigmentation pre and post PLE using the following"
  1. Investigator Global Assessment Scoring
  2. Diffuse Reflectance Spectroscopy
  3. Colorimetry
  4. Biopsy with melanocyte and melanin stains among other tissue markers
  5. Photography

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Middelkamp-Hup MA, Bos JD, Rius-Diaz F, Gonzalez S, Westerhof W. Treatment of vitiligo vulgaris with narrow-band UVB and oral Polypodium leucotomos extract: a randomized double-blind placebo-controlled study. J Eur Acad Dermatol Venereol. 2007 Aug;21(7):942-50. doi: 10.1111/j.1468-3083.2006.02132.x. PMID 17659004
- [Background] Middelkamp-Hup MA, Pathak MA, Parrado C, Goukassian D, Rius-Diaz F, Mihm MC, Fitzpatrick TB, Gonzalez S. Oral Polypodium leucotomos extract decreases ultraviolet-induced damage of human skin. J Am Acad Dermatol. 2004 Dec;51(6):910-8. doi: 10.1016/j.jaad.2004.06.027. PMID 15583582
- [Background] Mahmoud BH, Hexsel CL, Hamzavi IH, Lim HW. Effects of visible light on the skin. Photochem Photobiol. 2008 Mar-Apr;84(2):450-62. doi: 10.1111/j.1751-1097.2007.00286.x. Epub 2008 Jan 29. PMID 18248499
- [Background] Kollias N, Baqer A. An experimental study of the changes in pigmentation in human skin in vivo with visible and near infrared light. Photochem Photobiol. 1984 May;39(5):651-9. doi: 10.1111/j.1751-1097.1984.tb03905.x. No abstract available. PMID 6739557
- [Background] Porges SB, Kaidbey KH, Grove GL. Quantification of visible light-induced melanogenesis in human skin. Photodermatol. 1988 Oct;5(5):197-200. PMID 3222167
- [Background] Mahmoud BH, Ruvolo E, Hexsel CL, Liu Y, Owen MR, Kollias N, Lim HW, Hamzavi IH. Impact of long-wavelength UVA and visible light on melanocompetent skin. J Invest Dermatol. 2010 Aug;130(8):2092-7. doi: 10.1038/jid.2010.95. Epub 2010 Apr 22. PMID 20410914
- [Background] Hamanaka H, Miyachi Y, Imamura S. Photoprotective effect of topically applied superoxide dismutase on sunburn reaction in comparison with sunscreen. J Dermatol. 1990 Oct;17(10):595-8. doi: 10.1111/j.1346-8138.1990.tb01702.x. PMID 2273160
- [Derived] Mohammad TF, Kohli I, Nicholson CL, Treyger G, Chaowattanapanit S, Nahhas AF, Braunberger TL, Lim HW, Hamzavi IH. Oral Polypodium Leucotomos Extract and Its Impact on Visible Light-Induced Pigmentation in Human Subjects. J Drugs Dermatol. 2019 Dec 1;18(12):1198-1203. PMID 31859468